CLINICAL TRIAL: NCT05090761
Title: Is Serratus Anterior Plane Block (SAPB) With Adjuvant Medications Better at Managing Post-operative Pain Than Serratus Anterior Plane Block With Bupivacaine Alone in Patients Undergoing Video-assisted Thoracoscopy?
Brief Title: Serratus Anterior Plane Block With and Without Adjuvants in Video-assisted Thoracoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Sandeep Krishnan, Associate Professor of Anesthesiology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SAPB in thoracoscopy
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Post Operative Pain, Acute
Keywords: Serratus anterior plane block, video-assisted thoracoscopy, opioid consumption, magnesium, buprenorphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Magnesium Sulfate; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAPB (Active Comparator): 40 Patients - Patients will receive 30 mL of 0.25% bupivacaine injected below the serratus anterior muscle in the caudal direction using ultrasound guidance.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- SAPB with Mg (Active Comparator): 40 Patients - Patients will receive 30 mL of 0.25% bupivacaine with 150 mg of Mg injected below the serratus anterior muscle in the caudal direction using ultrasound guidance.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 150 mg
- SAPB with Mg and Buprenorphine (Active Comparator): 40 Patients - Patients will receive 30 mL of 0.25% bupivacaine with 150 mg of Mg and 300 mcg of buprenorphine injected below the serratus anterior muscle in the caudal direction using ultrasound guidance.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 150 mg, Buprenorphine 300 mcg

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Injection of Bupivacaine 0.25% Injectable Solution for SAPB
  Arms: SAPB
Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 150 mg — Injection of Bupivacaine 0.25% Injectable Solution for SAPB Addition of 150 mg of Magnesium Sulfate as adjuvant
  Arms: SAPB with Mg
Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 150 mg, Buprenorphine 300 mcg — Injection of Bupivacaine 0.25% Injectable Solution for SAPB Addition of 150 mg of Magnesium Sulfate and 300mcg Buprenorphine as adjuvants
  Arms: SAPB with Mg and Buprenorphine

SUMMARY:
The purpose of this study is to determine whether the addition of the serratus anterior plane block (SAPB) alone (30 mL of 0.25% bupivacaine) or plus Magnesium (150 mg of magnesium sulfate) or plus Magnesium + Buprenorphine (300 mcg) as adjuvants can improve post-operative pain in patients undergoing video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Many thoracic surgeons have switched from open thoracotomy to video-assisted thoracoscopy (VATS), when possible, in efforts to decrease length of hospital stays, decrease analgesic requirements, and decrease postoperative pain.

The serratus anterior plane block (SAPB) has been used effectively for the management of pain in the context of rib fractures, rib contusions, thoracoscopic surgery, thoracotomy, breast surgery, and post-mastectomy pain syndrome. It has been shown to have similar efficacy to thoracic epidurals in open thoracotomy.

The serratus anterior muscle originates from the anterior aspect of ribs 1 through 7-10 and inserts on the medial border of the scapula. It consists of 7 to 10 serrated tendinous projections that originate on each rib and is innervated by the long thoracic nerve. Deep and superficial potential spaces bound the serratus anterior. At the level of the fifth rib, the superficial plane forms from the anterior aspect of the serratus anterior and the posterior aspect of the latissimus dorsi muscle. The deep plane forms from the posterior aspect of the serratus anterior and the external intercostal muscles and ribs. Injecting in either plane will achieve analgesia to the anterolateral chest wall with reportedly similar efficacy and an equivalent area of cutaneous sensory loss.

The SAPB targets the lateral cutaneous branches of the thoracic intercostal nerves, which arise from the anterior rami of the thoracic spinal nerves and run in a neurovascular bundle immediately inferior to each rib. At the midaxillary line, the lateral cutaneous branches of the thoracic intercostal nerve traverse through the internal intercostal, external intercostal, and serratus anterior muscles innervating the musculature of the lateral thorax. These branches of the intercostal nerves, therefore, travel through the two potential spaces described above. Local anesthetic inserted into these planes will spread throughout the lateral chest wall, resulting in paresthesia of the T2 through T9 dermatomes of the anterolateral thorax.

Rebound pain is possible after serratus anterior block because analgesia provided by bupivacaine typically lasts around six hours. Local anesthetic systemic toxicity is a potential complication of regional anesthesia as well. For this reason, dilute anesthetic is used, and a maximum dose of 2 mg/kg of bupivacaine is the recommendation. Pneumothorax is a potential complication but would entail catastrophic error because the fascial planes targeted in this block are superficial to the ribs, and the pleural line can be visualized clearly on ultrasound. If a pneumothorax is suspected, ultrasound can help to confirm lung sliding immediately after the procedure. Nerve injury is unlikely given the needle is not steered directly at nerves, but instead towards the plane through which the nerves run.

The duration of traditional amide-based and ester-based regional anesthesia is normally limited to only a few hours as mentioned above. Techniques including continuous catheter placement or serial injections can be used to enhance the duration and effect of regional anesthesia for postoperative pain control. But these approaches can increase the risk of infection, toxicity, and cost. Therefore, alternative methods of extending the clinical duration of nerve blocks have been a topic of significant interest.

At SJMO patients who undergo a thoracoscopic procedures currently receive parenteral opioids or thoracic epidurals for management of pain.

The purpose of this study is to determine whether SAPB with bupivacaine and adjuvants can provide superior pain management (decrease pain scores) and decrease opioid consumption, without increasing nausea/vomiting, compared to patients receiving SAPB with bupivacaine alone in patients undergoing video-assisted thoracoscopy.

We will be assessing whether the addition of magnesium and buprenorphine to bupivacaine in SAPB will decrease visual analog scale (VAS) pain scores, reduce post-operative total opioid consumption (oral morphine equivalents), and decrease post-operative nausea and vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing video-assisted thoracoscopy

Exclusion Criteria:

* Patients with significant genetic or acquired clotting/bleeding disorders (hemophilia, DIC, etc.)
* Patients with significant platelet dysfunction
* Infection at site for regional anesthesia
* Allergy to local anesthetics
* Sepsis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative total opioid consumption (oral morphine equivalents) | 24 hours after surgery
  Total Opioid consumption 24 hours post surgery oral moral morphine equivalents
Visual analog scale (VAS) pain scores | 6 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain scores | 12 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain scores | 24 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)

SECONDARY OUTCOMES:
Incidence of post-operation nausea and vomiting (PONV) | 24 hours
  The percentage of the patients who had post-operative nausea and vomiting (PONV) within 24 hours of surgery
Acetaminophen consumption | 24 hours after surgery
  Total acetaminophen consumption in mg
NSAID (ketorolac) consumption | 24 hours after surgery
  Total NSAID consumption in mg

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Mercy Oakland Hospital, Pontiac, Michigan, United States

IPD SHARING:
Plan to Share IPD: No